CLINICAL TRIAL: NCT03792984
Title: The Effect of Calcium and Vitamin D Supplements as an Adjuvant Therapy to Metformin on Metabolic and Hormonal Disturbances in Polycystic Ovary Syndrome Patients
Brief Title: The Effect of Calcium and Vitamin D Supplements on Metabolic and Hormonal Disturbances in Polycystic Ovary Syndrome Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ph-CT-2685
Record Dates: First submitted 2018-12-18; First posted 2019-01-04 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2018-12

CONDITIONS: Polycystic Ovary Syndrome; Vitamin D Deficiency/Insufficiency
Keywords: Polycystic Ovary Syndrome; Calcium; Vitamin D; Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome; Vitamin D Deficiency | interventions — Cholecalciferol; Calcium Carbonate; Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin + Placebo (Placebo Comparator)
  Interventions: Drug: Metformin; Drug: Placebo
- Calcium carbonate + Vitamin D3 + Metformin (Experimental)
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Carbonate; Drug: Metformin

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 (Cholecalciferol) (6000 IU/daily). PO for 8 weeks.
  Arms: Calcium carbonate + Vitamin D3 + Metformin
Dietary Supplement: Calcium Carbonate — Calcium carbonate (1000 mg/daily). PO for 8 weeks.
  Arms: Calcium carbonate + Vitamin D3 + Metformin
Drug: Metformin — Metformin (1500 mg/daily; the metformin dose was increased stepwise, starting with 500 mg once daily for the 1st week, 500 mg twice daily in the 2nd week, followed by 500 mg 3 times daily from the 3rd week onward). PO for 8 weeks.
Drug: Placebo — PO for 8 weeks.
  Arms: Metformin + Placebo

SUMMARY:
The aim of this study is to investigate the safety and metabolic-hormonal efficiency of supplementation vitamin D deficient/insufficient PCOS women with (calcium +vitamin D + metformin) for 8 weeks compared to (placebo+ metformin).

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder among females of reproductive age. The main manifestations of this syndrome are ovulatory dysfunction, hyperandrogenism, and polycystic ovarian morphology. Noticeably, PCOS is associated with several metabolic disturbances such as insulin resistance, compensatory hyperinsulinemia, dyslipidemia and central obesity, which increase the risk for long-term complications like type 2 diabetes mellitus, metabolic syndrome, and cardiovascular diseases. Moreover, previous data demonstrated that, compared to normo-ovulatory women, PCOS patients might exhibit a dysregulation in the IGF system represented as an elevation in the serum levels of free Insulin-like growth factor-1 (IGF-1) and a reduction in the serum levels of Insulin-like growth factor binding protein-1 (IGFBP-1). However, the exact aetiology of PCOS remains unclear and current treatments are only moderately effective at controlling PCOS symptoms and preventing its complications. Growing evidence suggests a role of vitamin D in female reproductive diseases as the expression of Vitamin D Receptors (VDR) was identified in many organs throughout the female reproductive tract. On the top of that, vitamin D regulates over 300 genes, including genes that are important for glucose and lipid metabolism. Moreover, vitamin D deficiency is a common condition among women with PCOS, and several studies indicated an association between low levels of serum 25-hydroxyvitamin D (25-OH-Vitamin D) and manifestations of PCOS including insulin resistance, hyperandrogenism, and infertility. Further, a recent in-vitro study showed that vitamin D regulated steroidogenesis and IGFBP-1 production in cultured human ovarian cells, and many reports have suggested an interrelation between IGF-1 and vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* PCOS women aged 18-30 years diagnosed according to the Rotterdam criteria.
* Vitamin D deficiency or insufficiency according to the Endocrine Society Clinical Practice Guideline.
* Normal liver function.
* Normal kidney function.

Exclusion Criteria:

* Pregnant, postpartum or breastfeeding women.
* Females aged <18 or >30 years old.
* Patients who were diagnosed with androgen-secreting tumours, Cushing's syndrome, congenital adrenal hyperplasia, hyperprolactinemia, hypercalcemia, malabsorption disorders, diabetes mellitus, thyroid disorders, liver disease, renal disease, epilepsy, cardiovascular disease.
* History of kidney stones.
* Usage of any hormonal therapy, corticosteroids (other than topical corticosteroids forms), insulin sensitizers, hypolipidemic agents, anti-obesity medications, vitamin D or calcium supplements, anti-epileptic drugs, or any other drugs known to affect endocrine parameters, carbohydrate metabolism, or calciotropic hormone concentrations during the last 3 months.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Change in quantitative insulin sensitivity check index (QUICKI). | baseline, 8 weeks weeks.
  Assessment of QUICKI index at baseline and after 8 weeks of intervention.
Change in Raynaud's index. | baseline, 8 weeks weeks.
  Assessment of Raynaud's index at baseline and after 8 weeks of intervention.
Change in McAuley Index. | baseline, 8 weeks weeks.
  Assessment of McAuley Index at baseline and after 8 weeks of intervention.

SECONDARY OUTCOMES:
Change in glucose concentration. | baseline, 8 weeks.
  Assessment of serum concentration of glucose at baseline and after 8 weeks of intervention.
Change in insulin concentration. | baseline, 8 weeks.
  Assessment of serum concentration of insulin at baseline and after 8 weeks of intervention.
Change in homeostasis model assessment of insulin resistance index (HOMA-IR). | baseline, 8 weeks.
  Assessment of HOMA-IR index at baseline and after 8 weeks of intervention.
Change in homeostasis model assessment of β-cell function index (HOMA-B). | baseline, 8 weeks.
  Assessment of HOMA-B index at baseline and after 8 weeks of intervention.
Change in menstrual cycle abnormalities. | up to 8 weeks.
  Assessment of menstrual cycles regularity (having normal menstrual cycle 21-35 days) was done at baseline and during the study period using a calendar by recording the time of the onset of the menstrual periods and the duration of menses.
Change in hirsutism score | baseline, 8 weeks.
  Assessment of modified Ferriman-Gallwey score for hirsutism at baseline and after 8 weeks of intervention. (The score represents the hair growth in a male pattern on a woman shown in four different degrees of severity ( 0= no hair growth; 1= light hair growth; 2= moderate hair growth; 4= severe hair growth) in 9 different body parts; namely the upper lip, chin, chest, upper back, lower back, upper abdomen, lower abdomen, upper arms and thighs. The score is the sum of each region sub-score. Thus, it ranges between 0 and 36, where a score ≥ 6 was considered as a cut off Hirsutism).
Change in free testosterone concentration | baseline, 8 weeks.
  Assessment of serum free testosterone concentration at baseline and after 8 weeks of intervention.
Change in serum concentration of follicle-stimulating hormone (FSH) | baseline, 8 weeks or the next spontaneous menstrual cycle depending on menstrual cycle status.
  Assessment of serum concentration of FSH during the early follicular phase of menses at baseline and after 8 weeks of intervention if menstrual cycle regularity was reached during treatment period, or at baseline and the next spontaneous menstrual cycle after finishing the treatment if menstrual cycle regularity was not reached during treatment period.
Change in serum concentration of luteinizing hormone (LH) . | baseline, 8 weeks or the next spontaneous menstrual cycle depending on menstrual cycle status.
  Assessment of serum concentration of LH during the early follicular phase of menses at baseline and after 8 weeks of intervention if menstrual cycle regularity was reached during treatment period, or at baseline and the next spontaneous menstrual cycle after finishing the treatment if menstrual cycle regularity was not reached during treatment period.
Change in serum concentration of Insulin-like growth factor-1 (IGF-1). | baseline, 8 weeks.
  Assessment of serum concentration of IGF-1 at baseline and after 8 weeks of intervention.
Change in serum concentration of Insulin-like growth factor binding protein-1 (IGFBP-1). | baseline, 8 weeks.
  Assessment of serum concentration of IGFBP-1 at baseline and after 8 weeks of intervention.
Change in IGF-1 to IGFBP-1 ratio. | baseline, 8 weeks.
  Assessment of serum concentration of IGF-1 to IGFBP-1 ratio at baseline and after 8 weeks of intervention.
Change in lipid profile. | baseline, 8 weeks.
  Assessment of serum concentration of total cholesterol (TC), high-density lipoprotein cholesterol (HDL), low-density lipoprotein cholesterol (LDL), triglyceride (TG) and non-HDL cholesterol (non-HDL) at baseline and after 8 weeks of intervention.
Change in serum concentration of C-reactive protein (CRP) | baseline, 8 weeks.
  Assessment of serum concentration of CRP at baseline and after 8 weeks of intervention.
Change in Body mass index (BMI). | baseline, 8 weeks.
  Assessment of weight and height in an overnight fasting status without shoes with light clothes at baseline and after 8 weeks of intervention. Weight and height will be combined to report BMI in kg/m^2.
Change in waist circumference. | baseline, 8 weeks.
  Assessment of waist circumference in an overnight fasting status without shoes with light clothes at baseline and after 8 weeks of intervention.
Change in Hip circumference. | baseline, 8 weeks.
  Assessment of Hip circumference in an overnight fasting status without shoes with light clothes at baseline and after 8 weeks of intervention.
Change in waist to hip ratio. | baseline, 8 weeks.
  Assessment of waist to hip ratio in an overnight fasting status without shoes with light clothes at baseline and after 8 weeks of intervention.
Change in calcium concentration. | baseline, 8 weeks.
  Assessment of serum concentration of calcium at baseline and after 8 weeks of intervention.
Change in 25-OH-vitamin D concentration. | baseline, 8 weeks.
  Assessment of serum concentration of 25-OH-vitamin D at baseline and after 8 weeks of intervention.
Change in phosphorus concentration. | baseline, 8 weeks.
  Assessment of serum concentration of phosphorus at baseline and after 8 weeks of intervention.
Change in alanine transaminase (ALT) concentration. | baseline, 8 weeks.
  Assessment of serum concentration of ALT at baseline and after 8 weeks of intervention.
Change in aspartate transaminase (AST) concentration. | baseline, 8 weeks.
  Assessment of serum concentration of AST at baseline and after 8 weeks of intervention.
Change in urea concentration. | baseline, 8 weeks.
  Assessment of serum concentration of urea at baseline and after 8 weeks of intervention.
Change in creatinine concentration. | baseline, 8 weeks.
  Assessment of serum concentration of creatinine at baseline and after 8 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Kadoura, B Pharm, MD, Principal Investigator — Department of Pharmaceutics and Pharmaceutical Technology, Faculty of Pharmacy, Damascus University, Damascus, Syria; Abdul Hakim Nattouf, MD, PhD, Study Director — Professor at Department of Pharmaceutics and Pharmaceutical Technology, Faculty of Pharmacy, Damascus University, Damascus, Syria; Marwan Alhalabi, MD, PhD, Study Director — Professor at Department of Embryology and Reproductive Medicine, Faculty of Medicine, Damascus University, Damascus, Syria.
Locations (2):
- Syria (2):
  - Damascus University of Obstetrics and Gynecology Hospital, Damascus
  - Orient Hospital, Damascus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ameri P, Giusti A, Boschetti M, Murialdo G, Minuto F, Ferone D. Interactions between vitamin D and IGF-I: from physiology to clinical practice. Clin Endocrinol (Oxf). 2013 Oct;79(4):457-63. doi: 10.1111/cen.12268. Epub 2013 Aug 9. PMID 23789983
- [Background] Hahn S, Haselhorst U, Tan S, Quadbeck B, Schmidt M, Roesler S, Kimmig R, Mann K, Janssen OE. Low serum 25-hydroxyvitamin D concentrations are associated with insulin resistance and obesity in women with polycystic ovary syndrome. Exp Clin Endocrinol Diabetes. 2006 Nov;114(10):577-83. doi: 10.1055/s-2006-948308. PMID 17177140
- [Background] Irani M, Merhi Z. Role of vitamin D in ovarian physiology and its implication in reproduction: a systematic review. Fertil Steril. 2014 Aug;102(2):460-468.e3. doi: 10.1016/j.fertnstert.2014.04.046. Epub 2014 Jun 3. PMID 24933120
- [Background] Krul-Poel YH, Snackey C, Louwers Y, Lips P, Lambalk CB, Laven JS, Simsek S. The role of vitamin D in metabolic disturbances in polycystic ovary syndrome: a systematic review. Eur J Endocrinol. 2013 Oct 23;169(6):853-65. doi: 10.1530/EJE-13-0617. Print 2013 Dec. PMID 24044903
- [Background] Li HW, Brereton RE, Anderson RA, Wallace AM, Ho CK. Vitamin D deficiency is common and associated with metabolic risk factors in patients with polycystic ovary syndrome. Metabolism. 2011 Oct;60(10):1475-81. doi: 10.1016/j.metabol.2011.03.002. Epub 2011 May 6. PMID 21550088
- [Background] Ott J, Wattar L, Kurz C, Seemann R, Huber JC, Mayerhofer K, Vytiska-Binstorfer E. Parameters for calcium metabolism in women with polycystic ovary syndrome who undergo clomiphene citrate stimulation: a prospective cohort study. Eur J Endocrinol. 2012 May;166(5):897-902. doi: 10.1530/EJE-11-1070. Epub 2012 Feb 13. PMID 22330149
- [Background] Pal L, Zhang H, Williams J, Santoro NF, Diamond MP, Schlaff WD, Coutifaris C, Carson SA, Steinkampf MP, Carr BR, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Myers E, Legro RS; Reproductive Medicine Network. Vitamin D Status Relates to Reproductive Outcome in Women With Polycystic Ovary Syndrome: Secondary Analysis of a Multicenter Randomized Controlled Trial. J Clin Endocrinol Metab. 2016 Aug;101(8):3027-35. doi: 10.1210/jc.2015-4352. Epub 2016 May 17. PMID 27186859
- [Background] Parikh G, Varadinova M, Suwandhi P, Araki T, Rosenwaks Z, Poretsky L, Seto-Young D. Vitamin D regulates steroidogenesis and insulin-like growth factor binding protein-1 (IGFBP-1) production in human ovarian cells. Horm Metab Res. 2010 Sep;42(10):754-7. doi: 10.1055/s-0030-1262837. Epub 2010 Aug 13. PMID 20711952
- [Background] Thierry van Dessel HJ, Lee PD, Faessen G, Fauser BC, Giudice LC. Elevated serum levels of free insulin-like growth factor I in polycystic ovary syndrome. J Clin Endocrinol Metab. 1999 Sep;84(9):3030-5. doi: 10.1210/jcem.84.9.5941. PMID 10487660
- [Derived] Kadoura S, Alhalabi M, Nattouf AH. Effect of Calcium and Vitamin D Supplements as an Adjuvant Therapy to Metformin on Menstrual Cycle Abnormalities, Hormonal Profile, and IGF-1 System in Polycystic Ovary Syndrome Patients: A Randomized, Placebo-Controlled Clinical Trial. Adv Pharmacol Sci. 2019 Jul 1;2019:9680390. doi: 10.1155/2019/9680390. eCollection 2019. PMID 31354810